CLINICAL TRIAL: NCT03467763
Title: Trial of an Intervention to Improve Metformin Persistence and Adherence
Acronym: TreatMet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1706018342; K08HS023898 (AHRQ)
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Metformin Adverse Reaction; Tolerance

STUDY DESIGN:
Intervention Model Description: This study is an N-of-1 trial design that will recruit 20 previously metformin-intolerant patients for re-challenge with metformin in a double-blind scenario. Patients will be assigned to take their baseline medication regimen plus 2 weeks of 250 mg per day of metformin extended release, followed by 500 mg metformin XR, 750 mg, and 1,000 mg metformin XR with each treatment period separated by a 2-week course of placebo. Initial treatment, placebo or metformin XR, will be decided randomly.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, care providers, and investigators will be masked to the identity of the trial medication until the conclusion of the trial, and unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin Hydrochloride Extended Release (Active Comparator): Patients will be assigned to take their baseline medication regimen plus 2 weeks of 250 mg per day of metformin extended release, followed by 500 mg metformin XR, 750 mg, and 1,000 mg metformin XR with each treatment period separated by a 2-week course of placebo.
  Interventions: Drug: Metformin Extended Release Oral Tablet
- Placebo (Placebo Comparator): Patients will be assigned to take their baseline medication regimen plus 2 weeks of 250 mg per day of placebo, followed by 500 mg placebo, 750 mg, and 1,000 mg placebo with each treatment period separated by a 2-week course of metformin XR in the same increments of dosage.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — Metformin hydrochloride extended release tablets in dosages of 250 mg, 500 mg, 750 mg, and 1,000 mg. Individual encapsulations of metformin will contain dosages of 250 mg or 500 mg.
  Arms: Metformin Hydrochloride Extended Release
Drug: Placebo oral capsule — Placebo capsule
  Arms: Placebo

SUMMARY:
Metformin is a safe and effective first-line drug for type 2 diabetes that is also widely recommended for weight loss and diabetes prevention. But, metformin is associated with gastrointestinal and other side effects which prevent its use in 10-20% of patients and appear to limit the usable dose in others. This study is an N-of-1 trial design that will recruit 20 previously metformin-intolerant patients for re-challenge with metformin in a double-blind scenario. In this setting, 'intolerant' means either unable to take metformin at all, or unable to increase the dose past 1,000 mg despite the treating physician's recommendation to do so. Patients will be assigned to take their baseline medication regimen plus 2 weeks of 250 mg per day of metformin extended release, followed by 500 mg metformin XR, 750 mg, and 1,000 mg metformin XR with each treatment period separated by a 2-week course of placebo. Initial treatment, placebo or metformin XR, will be decided randomly. At the end of each two-week treatment period, participants will complete questionnaires assessing overall satisfaction with the medication, gastrointestinal symptoms, and adherence. Six months after the conclusion of the intervention, patients will be asked if they are continuing metformin at a higher dose than upon entry to the trial. This trial has two aims. First, to test the hypothesis that medication satisfaction will be the same during periods of placebo treatment and during periods of treatment with the active drug. The second aim is to test the hypothesis that > 30% of metformin-intolerant patients in an N of 1 crossover trial are able to tolerate higher-dose metformin at 6-months.

DETAILED DESCRIPTION:
Results have been presented in a single study arm as the order in which patients received drug or placebo was unique for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes, pre-diabetes, or obesity
* Previously attempted to take metformin for an above indication
* History of metformin intolerance (defined based on treating physician's assessment that a history of metformin intolerance (defined as the inability, due to side effects, to use metformin at the otherwise medically appropriate dose) exists, confirmed by the patient's recollection of the same history)

Exclusion Criteria:

* Contraindication to metformin (i.e, advanced renal or liver disease, history of metformin attributed lactic acidosis, or advanced heart failure)
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Igel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that results have been presented in a single study arm as the order in which participants received drug or placebo was unique for many patients, so that reporting a separate arm for each sequence of drug and placebo exposure would have resulted in reporting individual level results, potentially compromising patient confidentiality.
Groups:
- Metformin Hydrochloride Extended Release and Placebo: Participants took their baseline medication plus escalating doses of metformin in 250 mg increments, alternating with placebo in a randomized, double-blinded fashion.
  Patients were assigned to take their baseline medication regimen plus 2 weeks of 250 mg per day of metformin extended release, followed by 500 mg metformin XR, 750 mg, and 1,000 mg metformin XR with each treatment period separated by a 2-week course of placebo.
  Metformin Extended Release Oral Tablet: Metformin hydrochloride extended release tablets in dosages of 250 mg, 500 mg, 750 mg, and 1,000 mg. Individual encapsulations of metformin will contain dosages of 250 mg or 500 mg.
  Patients were assigned to take their baseline medication regimen plus 2 weeks of 250 mg per day of placebo, followed by 500 mg placebo, 750 mg, and 1,000 mg placebo with each treatment period separated by a 2-week course of metformin XR in the same increments of dosage.
  Placebo oral capsule: Placebo capsule
Period: Overall Study
Arm/Group | Metformin Hydrochloride Extended Release and Placebo
Started | 13
Weeks 1-2 | 13
Weeks 3-4 | 10
Weeks 5-6 | 8
Weeks 7-8 | 7
Weeks 9 - 10 | 6
Week 11-12 | 6
Weeks 13-14 | 2
Weeks 15-16 | 2
Completed (Subjects who stopped medication after completing a period are considered to have completed the study) | 10
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Please note that results have been presented in a single study arm as the order in which participants received drug or placebo was unique for many patients, so that reporting a separate arm for each sequence of drug and placebo exposure would have resulted in reporting individual level results, potentially compromising patient confidentiality.
Arm/Group | Metformin Hydrochloride Extended Release and Placebo
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black | 2
  White | 6
  Unknown or Not Reported | 3
  More Than One Race | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction as Measured by the Treatment Satisfaction Questionnaire for Medication (TSQM II)
Description: The primary outcome of this portion of the study will be the global satisfaction subscale of the Treatment Satisfaction Questionnaire for Medication (TSMQ II). The TSQM II is a 12-question survey with four satisfaction domains: effectiveness, side effects, convenience and global satisfaction. Each domain is described by a single numeric score. For each of these domains the lowest possible score (less satisfaction, ie a worse outcome) is 0, the highest (more satisfaction, ie a better outcome) is 100. We report this score global satisfaction domain (ie, subscale). (Note that the global satisfaction score is not a synthesis of the various subscales associated with each domain. It is a subscale in its own right comprised of distinct questions.)
Time Frame: 4-months
Population: The results from 3 participants were not analyzed as these participants were lost to follow-up or violated study protocol. Results are presented in two study arms, as reporting a separate arm for each sequence of drug and placebo exposure would have resulted in reporting individual level results, potentially compromising patient confidentiality. All patients contributed data to both arms except for 2 patients who had missing data during their placebo-exposed time.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Metformin Hydrochloride Extended Release: Metformin Extended Release Oral Tablet: Metformin hydrochloride extended release tablets in dosages of 250 mg, 500 mg, 750 mg, and 1,000 mg.
  Participants took their baseline medication plus escalating doses of metformin in 250 mg increments, alternating with placebo in a randomized, double-blinded fashion. The resulting regimen was 2 weeks of 250 mg per day of metformin extended release, followed by 500 mg metformin XR, 750 mg, and 1,000 mg metformin XR with each treatment period separated by a 2-week course of placebo.
  This arm includes only the person-time exposed to metformin XR.
- Placebo: Metformin Extended Release Oral Tablet: Metformin hydrochloride extended release tablets in dosages of 250 mg, 500 mg, 750 mg, and 1,000 mg.
  Participants took their baseline medication plus escalating doses of metformin in 250 mg increments, alternating with placebo in a randomized, double-blinded fashion. The resulting regimen was 2 weeks of 250 mg per day of metformin extended release, followed by 500 mg metformin XR, 750 mg, and 1,000 mg metformin XR with each treatment period separated by a 2-week course of placebo.
  This arm includes only the person-time exposed to placebo.
Arm/Group | Metformin Hydrochloride Extended Release | Placebo
Number analyzed (Participants) | 10 | 8
score on a scale | 39.42 (5.09) | 51.92 (4.57)

2. Primary Outcome: Number of Subjects Able to Tolerate Higher Dose of Metformin,
Description: For aim 2 of this study, the primary objective is to test the hypothesis > 30% of the patients enrolled in this study are able to tolerate (continue taking) a higher-dose of metformin at 6 months than they were taking at baseline.
Time Frame: 6-months
Population: Results from 3 participants not analyzed as these participants were lost to follow-up or violated study protocol. Results are presented in a single study arm, as reporting a separate arm for each sequence of drug and placebo exposure would have resulted in reporting individual level results, and because this outcome occurs only once per patient after the end of all placebo and metformin exposure periods it could not reported as two arms (placebo versus metformin.)
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin Hydrochloride Extended Release and Placebo
Number analyzed (Participants) | 10
Participants | 2

3. Secondary Outcome: Change in Score of Gastrointestinal Symptom Rating Scale (GSRS)
Description: For aim 1, the secondary objectives are to test the hypotheses that scores on a gastrointestinal symptom questionnaire are the same between between placebo and intervention periods; that adherence is the same between periods; and that the answer to the question 'Were you taking placebo or metformin for the past two weeks' is correct no more often than would be predicted by chance. Each question in the Gastrointestinal Symptom Rating Scale (GSRS) is scored on scale from 1 to 7 with 1 being no discomfort at all and 7 being very severe discomfort. The GSRS has separate questions to separately assess each of a range of potential GI symptoms (abdominal pain, reflux, diarrhoea, indigestion and constipation). Each symptom area can be described with the mean score of its contributing questions (so that the range in each symptom area is also 1 to 7, with lower numbers being better)
Time Frame: Reoccurring every 2-weeks for 4-months
Population: The results from 3 participants were not analyzed as these participants were lost to follow-up or violated study protocol. Results are presented in two study arms, as reporting a separate arm for each sequence of drug and placebo exposure would have resulted in reporting individual level results, potentially compromising patient confidentiality. All patients contributed data to both arms.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Metformin Hydrochloride Extended Release | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Reflux | 1.885 (0.24) | 1.78 (0.23)
  Diarrhea | 2.564 (0.29) | 2.346 (0.26)
  Constipation | 2.705 (0.23) | 2.667 (0.28)
  Abdominal Pain | 2.308 (0.21) | 2.346 (0.17)
  Indigestion | 2.50 (0.19) | 2.296 (0.26)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of active study participation, a maximum of 4 months for each patient.
Description: Results are presented in one study arm, as reporting a separate arm for each sequence of drug and placebo exposure would have resulted in reporting individual level results, potentially compromising patient confidentiality.
Arm/Group | Metformin Hydrochloride Extended Release and Placebo
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT03467763/Prot_SAP_000.pdf